CLINICAL TRIAL: NCT01427998
Title: A Phase Three Clinical Intervention Trial of Olive Leaves and Their Extracts in Human Diabetic Subjects
Brief Title: Effect of Olive Leaves as Hypoglycemic Agents in Diabetic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Diabetes, Director, Diabetes Unit, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WMC1111
Record Dates: First submitted 2011-08-03; First posted 2011-09-02 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes
Keywords: diabetes; blood glucose; olive leaf extract
MeSH Terms: conditions — Diabetes Mellitus | interventions — olive leaf extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- olive leaf extract (Active Comparator): Olive leaf polyphenol concentrate (OLPC) extraction OLPC was prepared from olive leaves as follows (Zaslave et al, 2005) : The leaves were randomly picked from the Barnea cultivar in the Jezreel Valley region of Israel and immediately freeze-dried on dry ice. After the leaves were thoroughly rinsed with sterile distilled water to remove dust, insecticides, and contaminating material, the leaves were ground and successively Soxhlet extracted with hexane for 3 h and 80% aqueous ethanol for 6 h. The alcoholic extract was concentrated under reduced pressure at 25 °C, and reconstituted with 30% ethanol in water.
  Interventions: Dietary Supplement: olive leaf extract
- placebo (Placebo Comparator): matched placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: olive leaf extract — olive leaf extract, 1 pill daily, 500 mg, for a duration of 14 wks
  Other Names: Olife
  Arms: olive leaf extract
Other: placebo — placebo
  Arms: placebo

SUMMARY:
Background: Animal studies indicate that olive leaf extract normalizes blood glucose. We hypothesized that olive leaf extract might be of benefit in human subjects.

Methods: A total of 79 adults with diabetes were randomly assigned to treatment with olive leaf extract capsules or matched placebo. Measures of glucose homeostasis including glucose, insulin and HbA1c were measured and compared by treatment group.

DETAILED DESCRIPTION:
The present study is a randomized, double blind, placebo controlled, clinical trial with a 14 week duration. Patients were randomized to treatment with a tablet of olive leaves or matching placebo in 1:1 ratio.

Patients were instructed to consume a diet consistent with ADA recommendations and an exercise training program was prescribed.

Weight, height, systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured in all subjects at the beginning and at the end of the study. Venous blood samples were drawn after an overnight fast of not less than 12 hours. Laboratory tests included fasting blood glucose (FBG), HbA1c, insulin, lipid panel and liver and renal function.

A total of 79 subjects (51 men, 28 women) aged 18-79 years with type 2 diabetes mellitus, were recruited from and followed up at an outpatient clinic. The subjects were selected from a series of 93 consecutive diabetic patients. Eligible patients had been diagnosed with T2DM for at least 1 year.

Subjects were randomized to treatment with olive leaf extract pills (1 500 mg pill daily taken orally) or matching placebo. The intervention was prepared as follows: olive leaves were picked from the Barnea cultivar in the Jezreel Valley region of Israel and immediately freeze-dried on dry ice. After the leaves were thoroughly rinsed with sterile distilled water to remove dust, insecticides, and contaminating material, the leaves were ground and successively Soxhlet extracted with hexane for 3 h and 80% aqueous ethanol for 6 h. The alcoholic extract was concentrated under reduced pressure at 25 °C, and reconstituted with 30% ethanol in water.

Olive leaves or placebo tablet was taken once daily orally throughout the study. All subjects continue their stable treatment to diabetes.

Data were analyzed using SPSS v10.0 (SPSS Inc., Chicago, USA). Continuous data were described a mean ± standard deviation and compared by treatment assignment using the t-test for independent samples. Associations between continuous variables were described by calculating the Pearson's correlation coefficients. Nominal variables such as sex and treatment assignment are described using frequency counts and compared by treatment assignment using the chi square test (exact as appropriate). All tests are two-sided and considered significant at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* adults
* type 2 diabetes

Exclusion Criteria:

* type 1 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 1999-08; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Serum glucose | 14 weeks
  serum glucose

SECONDARY OUTCOMES:
Plasma insulin | 14 weeks
  Plasma insulin

CONTACTS AND LOCATIONS:
Overall Officials: Julio Wainstein, MD, Principal Investigator — E. Wolfson Medical Center